CLINICAL TRIAL: NCT01534364
Title: Effect of a Preoperative Calorie Restriction on Renal Function After Cardiac Surgery
Brief Title: Brief Title:Effect of a Preoperative Calorie Restriction on Renal Function After Cardiac Surgery
Acronym: CR_KCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Volker Burst, MD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001; 00003355 (Registry Identifier: DRKS)
Record Dates: First submitted 2012-01-30; First posted 2012-02-16 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; acute kidney injury; diet; caloric restriction; cardiac surgery; cardiothoracic surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Ad libitum alimentation
- calorie restriction (Other): Calorie Restriction to 60% of the calculated daily energy rate from day -7 until day -1 (included) pre-surgery day 0 corresponds to day of surgery)
  Interventions: Other: calorie restriction

INTERVENTIONS:
Other: calorie restriction — Calorie Restriction to 60% of the calculated daily energy rate from day -7 until day -1 (included) pre-surgery (day 0 corresponds to day of surgery)
  Other Names: calorie restriction with Fresubin energy fibre drink
  Arms: calorie restriction

SUMMARY:
The aim of this study is to assess the effect of a diet prior to cardiac surgery on the common postoperative decline of renal function. Until now, there is no known drug or procedure to preserve the kidneys from this impairment. Patients with a known kidney disease are especially at risk. A potential beneficial effect of a diet prior to surgery has been shown in investigations in mammals, therefore this study will investigate if a preoperative diet in patients with known kidney disease and scheduled heart surgery can attenuate or prevent a postoperative loss of kidney function.

DETAILED DESCRIPTION:
Patients with cardiothoracic surgery are at risk for postoperative acute renal failure which is associated with significant morbidity and mortality. There is no drug or procedure known to prevent this loss of renal function. Experimental data suggests, that a preoperative caloric restriction might provide kidney protection in this context. This clinical trial investigates if this phenomenon is also applicable in humans. Patients with a increased risk for a postoperative renal failure due to known chronic kidney disease are randomized in 2 groups. Patients of the diet group receive a calorie restriction to 60% of the calculated daily energy rate from day -7 until day -1 (included) pre-surgery (day 0 corresponds to day of surgery). Patients of the control group receive alimentation ad libitum.

Primary objective is the increase of serum creatinine in mg/dl 24 h after induction of ischemia ("cross clamping") in comparison to baseline value obtained in the morning of the day of surgery (day 0) in order to analyse if a preoperative calorie restriction as a preventive strategy leads to a attenuation of postoperative kidney injury. Hypothesis: A seven day calorie restriction reduces the increase of serum creatinine after cardiac surgery in patients with known chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older
2. Caucasian origin
3. Scheduled cardiothoracic operation with employment of cardio-pulmonary bypass and a lead time of 11 days minimum.
4. Indication for cardiac surgery is determined by the cardiothoracic specialist
5. Patient and/or legal guardian must be willing and able to give written informed consent
6. one of the following risk factors:

   1. serum creatinine >1,1 mg/dl in male and > 0,9 mg/dl in female
   2. type 2 diabetes
   3. peripheral artery occlusive disease
   4. heart failure with NYHA III-IV (ejection fraction < 50 %)
   5. combined CABG and heart valve surgery
   6. further surgery after CABG or heart valve surgery

Exclusion Criteria:

1. End-stage renal disease (patient on dialysis)
2. Indwelling kidney transplant
3. Malnutrition (BMI < 18,5 kg/m2)
4. Body weight < 46 kg in male and < 51 kg in female
5. BMI > 35 kg/m2 or body weight > 120 kg
6. Catabolic state (serum albumine < 25 g/l)
7. Diet within the previous 4 weeks
8. Inappetence
9. Weight loss > 1 kg within the previous 2 weeks, if not explained by use of diuretics
10. Hospital stay during the last 7 days prior to cardiac surgery
11. Consuming underlying disease
12. Uncontrolled local or systemic infection
13. Contraindication for enteral nutrition.
14. Known allergy against or incompatibility with ingredients of the employed formula-diet
15. Pregnancy or breast feeding
16. Participation in other interventional clinical trials.
17. Missing safe method of contraception or missing occurence of menopause (in female)
18. Professional or private relationship between subject and the investigators or dependence on the investigators.
19. Placement in an institution based on official orders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The Increase of serum creatinine in mg/dl 24 h after induction of ischemia ("cross clamping") in comparison to baseline value obtained in the morning of the day of surgery (day 0). | baseline and 24 hours after induction of ischemia

SECONDARY OUTCOMES:
Urine Neutrophil-Gelatinase associated Lipocalin (NGAL in µg/l) 8h after induction of ischemia in comparison to baseline value obtained in the morning of the day of surgery (day 0). | baseline and 8 hours after induction of ischemia
C-reactive Protein (CRP) 24h after induction of ischemia | baseline and 24 h after induction of ischemia
Leucocyte count 24h after induction of ischemia | baseline and 24h after induction of ischemia
Creatinkinase (CK) 24h after induction of ischemia | baseline and 24 h after induction of ischemia
Troponin T 24h after induction of ischemia | baseline and 24 h after induction of ischemia
Lactate dehydrogenase 24h after induction of ischemia | baseline and 24 h after ischemia
N-terminal pro brain natriuretic peptide (NT-ProBNP) 24h after induction of ischemia | baseline and 24 h after ischemia
Serum lactate 24h after induction of ischemia | baseline and 24 hours after ischemia
Maximum increase of serum creatinine within the first 48 h after induction of ischemia | baseline and 48 hours after ischemia
Necessity of renal replacement therapy during hospital stay | pt will be followed for the duration of hospital stay, an expected average of 10 days
In-hospital mortality | pt will be followed for the duration of hospital stay, an expected average of 10 days
Time until fit for discharge | Participants will be followed for the duration of hospital stay, an expected average of 10 days
Length of hospital stay | Pt will be followed for the duration of hospital stay an expected average of 10 days
Echocardiographic estimated left-ventricular ejection fraction as per file, if assessed postoperatively | baseline and postoperatively, expected within 10 days after operation
Occurrence of acute renal failure in accordance with KDIGO I, II, III | Patients will be followed during hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Grundmann F, Muller RU, Reppenhorst A, Hulswitt L, Spath MR, Kubacki T, Scherner M, Faust M, Becker I, Wahlers T, Schermer B, Benzing T, Burst V. Preoperative Short-Term Calorie Restriction for Prevention of Acute Kidney Injury After Cardiac Surgery: A Randomized, Controlled, Open-Label, Pilot Trial. J Am Heart Assoc. 2018 Mar 13;7(6):e008181. doi: 10.1161/JAHA.117.008181. PMID 29535139